CLINICAL TRIAL: NCT05682794
Title: Transanal Versus Laparoscopic Total Mesorectal Excision: a Prospective Observational Cohort
Brief Title: Transanal Versus Laparoscopic Total Mesorectal Excision: a Cohort
Status: Completed | Type: Observational
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Yanhong Deng, Professor, Sun Yat-sen University
Other Study IDs: GIHSYSU-32
Record Dates: First submitted 2022-12-27; First posted 2023-01-12 (Actual); Last update posted 2023-01-12 (Actual); Status verified 2022-12

CONDITIONS: Rectal Cancer
Keywords: Rectal cancer; taTME; Local recurrence
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- taTME: patients who underwent transanal total mesorectal excision
  Interventions: Procedure: transanal total mesorectal excision
- laTME: patients who underwent laparoscopic total mesorectal excision

INTERVENTIONS:
Procedure: transanal total mesorectal excision — transanal TME
  Other Names: laparoscopic total mesorectal excision
  Groups: taTME

SUMMARY:
The purpose of this study was to compare the long-term oncology outcomes and specimen quality of taTME and laTME in the treatment of middle and low rectal cancer by a large sample cohort. At the same time, the local recurrence following a primary rectal cancer resection was analyzed to respond to the concerns about the event of the national suspension for TaTME due to the high local recurrence rate in Norway.

DETAILED DESCRIPTION:
Laparoscopic surgery is considered to have better visualization for more accurate separation and further injury reduction than open surgery. However, the oncology outcomes are still controversial. Especially in the challenging patients who have narrow and deep pelvic, the disadvantage that it is difficult to obtain high-quality resected specimens during laparoscopic TME (laTME) surgery is considered to be magnified. It is considered transanal total mesorectal excision (taTME) is an alternative method to solve this "old problem". However, as a new technology that has been around for only 10 years, the applicability of taTME worldwide needs to be further proved in long-term oncology. This prospective cohort study aimed to compare taTME surgery to laTME surgery for mid and low-rectal cancer on long-term oncology outcomes from a single, experienced Chinese center that was an early adopter of taTME.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 and 80 years old
2. Confirmed rectal adenocarcinoma cancer pathologically
3. Tumor location ≦ 12 cm from the anal margin
4. Willing and able to provide written informed consent for participation in this study

Exclusion Criteria:

1. Distant metastasis before surgery
2. More than one colorectal tumor at diagnosis
3. Familial adenomatous polyposis
4. Recurrent rectal cancer
5. Undergo transanal minimally invasive surgery
6. Undergo palliative treatment
7. Undergo emergency surgery

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Low-mid rectal cancer within Stage III.
Sampling Method: Non-Probability Sample
Enrollment: 2502 (Actual)
Dates: Start 2014-01 (Actual); Primary Completion 2022-10 (Actual); Study Completion 2022-10 (Actual)

PRIMARY OUTCOMES:
Overall survival rate | 5 years after the surgery
disease-free survival ratev | 5 years after the surgery

SECONDARY OUTCOMES:
Local recurrence rate | 3 years after the surgery
  Local recurrence was defined as radiologic or histopathologic evidence of any recurrent disease deposit located in the pelvis in the prior area of dissection following a primary rectal cancer resection, with or without distal metastasis
Cancer special survival rate | 5 years after the surgery
  Cancer special survival was defined as the time from the date of primary rectal cancer resection to the date of death caused by rectal cancer.
Quality of the mesorectum specimen | 30 days after the surgery
  The quality of the resected mesorectum was classified into three grades: (a) incomplete, (b) nearly complete, and (c) complete
CRM status | 30 days after the surgery
  The CRM was regarded as positive if the tumor distance or malignant lymph node to CRM was ≦1 mm.
DRM status | 30 days after the surgery
  The DRM was regarded as positive if it was microscopically involved by or ≦1 mm from the tumor margins.

CONTACTS AND LOCATIONS:
Overall Officials: Liang Kang, Principal Investigator — Sun Yat-sen University

IPD SHARING:
Plan to Share IPD: Undecided
The data can be obtained with a proper request.

REFERENCES:
- [Derived] Li Z, Liu H, Luo S, Hou Y, Zhou Y, Zheng X, Zhang X, Huang L, Zeng Z, Kang L. Long-term oncological outcomes of transanal versus laparoscopic total mesorectal excision for mid-low rectal cancer: a retrospective analysis of 2502 patients. Int J Surg. 2024 Mar 1;110(3):1611-1619. doi: 10.1097/JS9.0000000000000992. PMID 38091943